CLINICAL TRIAL: NCT04187924
Title: Effects of the Addition of the SIMEOX Device on Autogenic Drainage in Patients With Cystic Fibrosis
Brief Title: Effects of SIMEOX on Airway Clearance in Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, William Poncin, PT, PhD, Principal Investigator, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SIMEOX-003
Record Dates: First submitted 2019-11-27; First posted 2019-12-05 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autogenic drainage (Active Comparator): Patients will have to perform a 30-min session of autogenic drainage. Sputum will be collected during the session.
  Interventions: Other: Autogenic drainage
- SIMEOX + Autogenic drainage (Active Comparator): Patients will have to perform a 30-min session of autogenic drainage with the SIMEOX device. Sputum will be collected during the session.
  Interventions: Device: SIMEOX + Autogenic drainage

INTERVENTIONS:
Other: Autogenic drainage — Autogenic drainage is an airway clearance technique characterised by breathing control using expiratory airflow to mobilise secretions from smaller to larger airways. The secretions will be collected during the physiotherapy session and during the 24 hours following the session.
  Arms: Autogenic drainage
Device: SIMEOX + Autogenic drainage — SIMEOX is a device generating a succession of gentle depression at the mouth during the expiratory phase associated with autogenic drainage.
  Arms: SIMEOX + Autogenic drainage

SUMMARY:
This study will investigate the contribution of SIMEOX technology on the effectiveness of bronchial drainage.

This is a crossover study to evaluate the contribution of SIMEOX on the effectiveness of bronchial drainage (verified by the amount of sputum secretions, the rheology of sputum secretions and the subjective sensation of ease of sputum) in patients with cystic fibrosis.

Patients will perform, in randomized order (1) a 30-min session of autogenic drainage, (2) a 30-min session of autogenic drainage with the SIMEOX device. Sputum will be collected during and after the session. The two sessions will be performed with minimum washout time of 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Adults with cystic fibrosis
* Chronic bronchorrhea, able to expectorate by themselves
* Hospitalized

Exclusion Criteria:

* Regular use of SIMEOX,
* Difficulties in understanding instructions,
* Severe cardiac comorbidity.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-11-27 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Amount of sputum secretion | 30-min
  Total wet weight and dry weight of sputum collected in the 24-h following each intervention will be quantified.
Mucus viscoelasticity | 30-min
  Change in rheological properties of the sputum before and after each intervention will be analyzed using a rheometer. We will use the Rheomuco (Rheonova) reometer to obtain the differences in elasticity (G'), viscosity (G')' and elastic modulus ratio (tanδ) of the secretions collected before and after each intervention.
Subjective feeling of ease to expectorate | 3-min
  A Visual Analogue Scale (VAS) will be used to measure subjective feeling of ease of expectoration during each intervention.
  The visual analogue scale (VAS) is a semi-objective rating system that will be used to quantify the subjective feeling of ease to expectorate. The VAS is represented by a horizontal line marked 0 to 10, where "0" indicates "very easy to expectorate" and "10" indicates "not easy to expectorate at all". The lower the score, the easier it is to expectorate.

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No